CLINICAL TRIAL: NCT06735976
Title: Efficacy & Safety of LOBO™ Vascular Occlusion Device for Embolization of Pulmonary Arteriovenous Malformations (PAVM)
Brief Title: Efficacy & Safety of LOBO™ Vascular Occlusion Device for Embolization of Pulmonary Arteriovenous Malformations
Acronym: PAVM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Okami Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-2233
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arteriovenous Malformations
Keywords: Embolization; Pulmonary Arteriovenous Malformations; PAVM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PAVM Embolization (Other): This study consists of one group. All participants will undergo PAVM embolization with a LOBO™ device.
  Interventions: Device: PAVM Embolization; Device: PAVM Embolization with a LOBO™ device

INTERVENTIONS:
Device: PAVM Embolization — This study consists of one group. All participants will undergo PAVM embolization with a LOBO™ device.
Device: PAVM Embolization with a LOBO™ device — Participants will undergo PAVM embolization with the LOBO™ device per standard of care.

SUMMARY:
The goal of this clinical trial is to evaluate both the technical success and efficacy of using the LOBO™ device in patients undergoing embolization of Pulmonary Arteriovenous Malformations (PAVM). The main question[s] it aims to answer [is/are]:

* What is the technical success rate, the number of LOBO™ devices needed for occlusion, and time to occlusion for each feeding artery during PAVM embolization using the LOBO™ device?
* What is the short-term occlusion rate of the LOBO™ device for PAVM embolization (6 months post-embolization)?
* What are the medium- and long-term occlusion rate of the LOBO™ device in PAVMs (12 months and 36 months post embolization)?

Researchers will compare the percentage of LOBO™ embolized PAVMs that develop recanalization at 6, 12, and 36- month intervals compared to percentage of conventionally embolized PAVMs that develop recanalization at the same intervals.

Participants will undergo the embolization procedure and be followed for 36 months after the procedure. There will be a total of 4 study visits:

* Treatment visit
* 6-Month Follow-up visit
* 12-Month Follow-up visit
* 36-Month Follow-up visit

At each clinical follow-up visit participants will undergo imaging with a computed tomography angiography (CTA) of the chest.

DETAILED DESCRIPTION:
This is a prospective, interventional, single-center investigation involving the enrollment of 30 participants with PAVMs with feeding arteries ≥2 mm in diameter. Per standard of care and current clinical practice at UNC, all patients are first evaluated at the UNC Hereditary Hemorrhagic Telangiectasia (HHT) clinic which is run by the UNC Hematology Division. Based on clinical symptoms and signs (shortness of breath, hypoxia, positive bubble study, history of stroke or transient ischemic attack), and/or imaging findings (i.e., feeding artery size) on chest computed tomography angiography (CTA), patients are referred to interventional radiology for consultation for PAVM embolization. At this time, patients will be approached for enrollment in this study. This study aims to assess the technical success and rates of recanalization of PAVMs embolized using the LOBO™ device.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 PAVM with a feeding artery ≥2 mm in diameter and a feeding artery amenable to the use of LOBO™ device (i.e. feeding artery length of ≥1 cm). Given the length of embolic devices including LOBO™, the proximal vessel length to the PAVM sac must be of sufficient size for embolization to be feasible. If patients have at least 1 PAVM where the feeding artery length is ≥1 cm, they are eligible for enrollment.
* Patients with multiple PAVMs meeting eligibility criteria may be enrolled with the intent of embolizing multiple different PAVMs with the LOBO™ device in the same embolization session or in separate sessions.
* Estimated Glomerular Filtration Rate >30 ml/min
* Per standard of care (SOC), all pregnant women to be enrolled must be in their 2nd or 3rd trimesters

Exclusion Criteria:

* Confounding bleeding disorders other than HHT
* Life-threatening iodinated contrast allergy not amenable to prophylactic therapy with steroids
* Underlying coagulopathy
* Patients on anti-platelets or anti-coagulation medications

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Technical Success | At treatment until stasis is achieved. Approximately 1 - 2 hours.
  Technical success will be defined as the successful deployment of the LOBO™ device in the intended vessel and complete occlusion of the vessel. Successful deployment will be defined as 1) no technical malfunctions in the LOBO™ deployment system that leads to an inability to deploy the device and 2) deployment of the device into the intended vessel and not into surrounding vessels. Complete occlusion will be defined as complete cessation of blood flow through the embolized vessel based on intraprocedural angiography.

SECONDARY OUTCOMES:
Mean Number of LOBO Plugs | At treatment until stasis is achieved. Approx. 1 - 2 hours.
  Descriptive statistics for the number of LOBO™ devices needed for technical success will be reported.
Mean Time to Complete Occlusion | At treatment until stasis is achieved. Approx. 1 - 2 hours.
  Descriptive statistics for the time to completion will be reported.
Short-term Occlusion Rate | 6 months post-embolization
  Recanalization will be defined as contrast visualization through the plug or the aneurysmal sac on follow-up CTA's. Interpretation of these images will be done by standard clinical radiologists and not research personnel. The reading radiologist's interpretation will be used to determine if recanalization has occurred.
Medium- and Long-term Occlusion Rates | 12 months and 36 months post-embolization
  Recanalization will be defined as contrast visualization through the plug or the aneurysmal sac on follow-up CTA's. Interpretation of these images will be done by standard clinical radiologists and not research personnel. The reading radiologist's interpretation will be used to determine if recanalization has occurred.
Recanalization Rates by Modality (LOBO vs conventional) | 6, 12, and 36-months post-embolization
  Proportion of LOBO™ embolized PAVMs that develop recanalization at 6, 12, and 36- month intervals compared to proportion of conventionally embolized PAVMs (those embolized with coils, Amplatzer, MVPs) that develop recanalization at the same intervals. The retrospective comparator group will consist of patients who have undergone conventional embolization at UNC in a separate trial.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Kokabi, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.